CLINICAL TRIAL: NCT05283915
Title: An Open-label Phase 1, Pharmacokinetic and Tolerability Study of Tolebrutinib Given as a Single Dose in Adult Participants With Mild Hepatic Impairment, and in Matched Participants With Normal Hepatic Function
Brief Title: Study to Assess the Plasma Concentration of Tolebrutinib Given as a Tablet to Adult Participants With Mild Hepatic Impairment Compared to Participants With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POP16398; U1111-1269-6849 (Registry Identifier: ICTRP); 2022-003098-47 (EudraCT Number)
Record Dates: First submitted 2022-03-07; First posted 2022-03-17 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Hepatic Function Abnormal
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mild hepatic impairment group (Experimental): Single dose of tolebrutinib (SAR442168) will be administered on Day 1 under fed condition
  Interventions: Drug: tolebrutinib
- Normal hepatic function group (Experimental): Single dose of tolebrutinib (SAR442168) will be administered on Day 1 under fed condition
  Interventions: Drug: tolebrutinib

INTERVENTIONS:
Drug: tolebrutinib — Pharmaceutical form: Film-coated tablet Route of administration: oral

SUMMARY:
The purpose of this parallel group, Phase 1, open-label, 2-arm, single dose, multi-center study is to assess the effect of mild hepatic impairment on pharmacokinetics (PK), safety and tolerability of tolebrutinib compared with normal hepatic function, in male and female participants aged 18 to 79 years.

DETAILED DESCRIPTION:
The total duration of the study per participant is up to 41 days including:

* A screening period of up to 4 weeks (Days -28 to -2)
* A 5-day, open-label treatment period
* Up to 7 days post-treatment follow-up period

ELIGIBILITY:
Inclusion Criteria:

For participants with mild hepatic impairment

* Stable chronic liver disease assessed by medical history, physical examination, and laboratory values
* Child-Pugh total score ranging from 5 to 6, inclusive.
* Laboratory parameters within the acceptable range for participants with hepatic impairment; however, estimated glomerular filtration rate (eGFR) should be above or equal to 60 mL/min

For all participants

* Body weight between 50.0 and 115.0 kg, inclusive, if male, between 40.0 and 100 kg, inclusive, if female, and body mass index (BMI) within the range 18 to 40 kg/m2, inclusive, at screening.
* Participant with platelet count ≥150 000/μL at the screening visit and at Day -1

Exclusion Criteria:

For all participants :

* Symptomatic postural hypotension, whatever the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥30 mmHg within 3 minutes when changing from supine to standing position at screening and Day -1
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only: more than twice a month).
* History of drug or alcohol abuse within 1 year before inclusion.
* Smoking regularly more than 15 cigarettes or equivalent per day, unable to refrain from smoking over 8 cigarettes per day during the institutionalization.
* Any consumption of citrus fruits (grapefruit, orange, etc) or their juices within 72 hours before inclusion.
* Use of any herbal medicines 2 weeks before IMP administration
* Treatment with a strong or moderate CYP3A inhibitors, a strong, moderate or mild CYP2C8 inhibitors OR CYP3A, CYP2C8 inducers within 14 days before the study treatment administration or 5 half-lives, whichever is longer

Specific for participants with mild hepatic impairment:

* Uncontrolled clinically relevant cardiovascular, pulmonary, gastrointestinal, metabolic, hematological, neurological, psychiatric, systemic, ocular, gynecologic, renal, infectious disease, moderate or severe hepatic impairment (Child-Pugh total score greater than or equal to 7), or signs of acute illness.
* Hepatocarcinoma.
* Acute liver disease.
* Hepatic encephalopathy Grade 2, 3, and 4.
* Esophageal bleeding which is caused by esophageal varices within 3 months before inclusion.

NOTE: Other Inclusion/Exclusion criteria may apply. The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Assessment of PK parameters Tolebrutinib: AUC | From Day 1 to Day 4
  Area under the plasma concentration (AUC) versus time curve extrapolated to infinity
Assessment of PK parameters M2: AUC | From Day 1 to Day 4

SECONDARY OUTCOMES:
Assessment of PK parameters Tolebrutinib: Cmax | From Day 1 to Day 4
  Maximum plasma concentration observed (Cmax)
Assessment of PK parameters M2: Cmax | From Day 1 to Day 4
Assessment of PK parameters Tolebrutinib: AUClast | From Day 1 to Day 4
  Area under the serum concentration versus time curve calculated using the trapezoidal method from time zero to the real time Tlast
Assessment of PK parameters M2: AUClast | From Day 1 to Day 4
Number of participants with treatment-emergent adverse events (TEAEs) | From Day 1 to Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami Site Number : 8400002, Miami, Florida
  - Nucleus Network Site Number : 8400001, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: POP16398 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25332&tenant=MT_SNY_9011